CLINICAL TRIAL: NCT01416623
Title: A Phase I Study of Henatinib in Patients With Advanced Solid Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNTN-I
Record Dates: First submitted 2011-08-12; First posted 2011-08-15 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Advanced Solid Cancer
Keywords: Advanced solid cancer; Henatinib; phase I
MeSH Terms: interventions — 2-((5-fluoro-1,2-dihydro-2-oxo-3H-indol-3-ylidene)methyl)-5-(2-hydroxy-3-morpholinopropyl)-3-methyl-5,6,7,8-tetrahydro-1H-pyrrolo(3,2-c)azepin-4-ketone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Henatinib (Experimental): Henatinib either at 12.5,25,37.5,50,62.5,75,87.5 or 100 mg, p.o. once daily
  Interventions: Drug: henatinib

INTERVENTIONS:
Drug: henatinib — Henatinib Maleate Tablets

SUMMARY:
Henatinib is a novel oral multitargeted tyrosine kinase inhibitor with antitumor and antiangiogenic activities. This study is designed to evaluate the safety and tolerability of Henatinib in patients with Advanced Solid Malignancies

DETAILED DESCRIPTION:
1. To evaluate the safety and tolerability of Henatinib, and the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT).
2. To determine the pharmacokinetic profile of Henatinib and its metabolites .
3. To assess preliminary antitumor activity .
4. To determine preliminary regimen for phase II study .

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologic (except sputum smear) confirmed metastatic or locally advanced solid tumor (At least one measurable lesion longest diameter ≥20 mm using conventional techniques or larger than 10 mm in diameter by spiral CT scan).
2. Life expectancy of more than 12 weeks.
3. Lack of standard treatment or standard treatment failure.
4. Screening laboratory values within the following parameters:

   1. HB:≥90g/L
   2. ANC:≥1.5×109/L
   3. PLT:≥100×109/L
5. ALT and AST:≤1.5×ULN(But if the liver metastases, ALT and AST:≤5×ULN) 1. Serum total bilirubin:≤1.5×ULN 2. Serum creatinine:≤1.5×ULN 3. Creatinie clearance rate:≥60ml/min 4. Electrolytes normal or return to normal after treatment
6. Recovery from all clinically significant AEs related to prior therapies. Duration from the latest therapy is more than 6 weeks for nitroso or mitomycin, or more than 4 weeks for radiotherapy, chemotherapy, immunotherapy or other anti-cancer treatments (such as testing drugs, biologics, hormones or surgery).
7. Signed and dated informed consent. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedure.

Exclusion Criteria:

1. Evidence of CNS metastasis.
2. Major surgery, open biopsy, or obvious trauma within 4 weeks before treatment.
3. Obvious peritoneal implantation or pelvic obstruction.
4. II level or above, peripheral neuropathy (NCI CTC AE v3.0).
5. Known history of neurological or psychiatric disease.
6. Suffering from high blood pressure and can not be reduced to the following range by monotherapy (systolic blood pressure <140 mmHg, diastolic blood pressure <90 mmHg).
7. History of heart disease:> NYHA II class congestive heart failure; unstable coronary artery disease (patients who had last myocardial infarction 12 months before can be enrolled), arrhythmias - requires antiarrhythmic drug therapy. Bazett's corrected QTc ≥ 480 ms or can not be measured. (Note: If ECG QTc interval ≥ 480 ms during the screening period, you must repeat 2 times, separated by at least 24 hours, the average QTc of the 3 times must be <480 s, the patient can be enrolled in this study) .
8. Coagulopathy (PT> 16 s, APTT> 43 s, TT> 21 s, Fbg <2 g / L), with a bleeding tendency or are receiving the therapy of thrombolysis or anticoagulation.
9. Confirmed active gastrointestinal ulcers.
10. Active severe infection (> NCI-CTC 3.0 standard 2).
11. Patients with severe epilepsy requires drug treatment (such as steroids or anti-epileptic drugs).
12. Other serious illness or condition.
13. Treated with VEGFR TKIs such as sunitinib or solafenib before study entry.
14. Less than 4 weeks from the last clinical trial.
15. Pregnancy, breast-feeding women or women of childbearing age without effective contraception.
16. Allergic or known history of hypersensitivity to henatinib or any of it components.
17. Drug abuse, the drug and mental illness may affect the patients participation in this study and the assessment of the research results.
18. Any unstable or likely situation that harms the safety and compliance of the patients in this study.
19. Any factors that influence the usage of oral administration.
20. Evidence of significant medical illness that in the investigator's judgment will substantially increase the risk associated with the subject's participation in and completion of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-09; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
The maximum-tolerated dose (MTD) regimen of henatinib will be defined as the maximum dose level at which no more than one subject out of six experiences a dose-limiting toxicity (DLT) after completing one treatment cycle. | 4 weeks

SECONDARY OUTCOMES:
Number of participants with adverse events | 8 weeks
Henatinib pharmacokinetic parameters may include AUC, Cmax, Tmax, and t1/2. | 4 weeks
Objective response rate (ORR) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: jin Li, Dr, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China